CLINICAL TRIAL: NCT06913140
Title: Preoperative Ultrasound Guided Thoracic Erector Spinae Plane Block Versus Costoclavicular Block for Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Naeem, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35844/9/22
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Preoperative; Ultrasound; Thoracic Erector Spinae Plane Block; Costoclavicular Block; Shoulder Arthroscopy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector Spinae plane Block group (Experimental): Patients received (20ml) plain bupivacaine 0.25% injected beneath the erector spinae muscle sheath at the level of the second thoracic segment (T2)
  Interventions: Drug: Erector Spinae plane Block
- Costoclavicular block group (Experimental): Patients received (20ml) plain bupivacaine 0.25% injected in the costoclavicular space lateral to axillary artery
  Interventions: Drug: Costoclavicular block
- Control group (Sham Comparator): Patients received sham block .
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Erector Spinae plane Block — Patients received (20ml) plain bupivacaine 0.25% injected beneath the erector spinae muscle sheath at the level of the second thoracic segment (T2)
  Other Names: Bupivacaine 0.25%
  Arms: Erector Spinae plane Block group
Drug: Costoclavicular block — Patients received (20ml) plain bupivacaine 0.25% injected in the costoclavicular space lateral to axillary artery.
  Other Names: Bupivacaine 0.25%
  Arms: Costoclavicular block group
Drug: Control group — Patients received sham block
  Other Names: Sham block
  Arms: Control group

SUMMARY:
This study was conducted to compare the perioperative analgesic effect of ultrasound guided high thoracic erector spinae plane block versus ultrasound guided costoclavicular block for shoulder arthroscopy

DETAILED DESCRIPTION:
Shoulder surgery is one of the most common orthopedic surgical procedures that causes severe pain . Pain management in such patients is very important because pain relief allows early mobilization, effective postoperative rehabilitation, and shorter hospitalization stays. Several regional anesthesia techniques have been used for pain management following shoulder surgery. Interscalene brachial plexus block (ISB) is the gold standard analgesic technique for shoulder procedures, but this method can lead to some serious complications, such as hemidiaphragmatic paralysis (HDP), Horner's syndrome, and hoarseness.

The costoclavicular block (CCB) was introduced as infraclavicular approach, first described in 2015 , targets the brachial plexus in the costoclavicular space where its three cords are tightly clustered together lateral to the axillary artery and more superficially than with the classical approach of infraclavicular fossa . Recently, Garcia-Vittoria et al have suggested that the costoclavicular space could also serve as a retrograde channel to supraclavicular brachial plexus blocks, so if local anesthetic (LA) injected in the costoclavicular space can reliably reach the supraclavicular brachial plexus enabling reliable anesthesia including anesthesia to the suprascapular nerve during shoulder surgery, one could achieve analgesic parity with small-volume supraclavicular block (and ISB) while retaining the 0% incidence of HDP seen with infraclavicular blocks.

Erector spinae plane block (ESPB) is a relatively novel block and was first described for chronic thoracic neuropathic pain in 2016 (. It is an interfascial plane block, but it may be classified as a paraspinal block due to its mechanism of action and injection site

ELIGIBILITY:
Inclusion Criteria:

* 90 patients admitted for elective unilateral shoulder arthroscopy.
* Aged (21 - 65) years.
* American Society of Anesthesiologists (ASA) physical activity I, II

Exclusion Criteria:

* Patient refusal.
* Patient with neurological deficit.
* Patient with bleeding disorders (coagulopathy, thrombocytopenia anticoagulant and antiplatelets drugs).
* Uncooperative patient.
* Infection at the block injection site.
* Patients with history of allergy to local anaesthetics

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Total Pethidine consumption | 24 hours postoperatively
  Each patient was instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable") at (T 30 min, 2, 4, 6,12, 18, 24 h, non-steroidal anti-inflammatory drugs were given (ketorolac 30mg) to all patient /8 h and if VAS > 4 intravenous pethidine 0.5 mg / kg per dose.

SECONDARY OUTCOMES:
Time to first analgesic request after surgery | 24 hours postoperatively
  Time to 1st request for the rescue of analgesia (time from the end of surgery till first dose of morphine administrated) was recorded.
Degree of pain | 24 hours postoperatively
  Each patient was instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable") at (T 30 min, 2, 4, 6,12, 18, 24 h, non-steroidal anti-inflammatory drugs were given (ketorolac 30mg) to all patient /8 h and if VAS > 4 intravenous pethidine 0.5 mg / kg per dose.
Complications | 24 hours postoperatively
  Complications (Hematoma, pneumothorax, persistent numbness/ paraesthesia or motor deficit one week after the surgery) were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author